CLINICAL TRIAL: NCT03240991
Title: Study of Clinical, Biological Characteristics and Quality of Life of Patients With Hereditary or Acquired Non Drug-induced Bradykinin-mediated Angioedema, Monitored in Besançon's Partner Site Reference Center for Studies of Kinin-mediated Angioedema (CREAK)
Acronym: QUALANGIO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: P/2016/302
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Angioedema
Keywords: bradykinin-mediated angiodema; quality of life
MeSH Terms: conditions — Angioedema | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Quality of life questionnaires: Data will be collected retrospectively and prospectively.
  Interventions: Other: Quality of life

INTERVENTIONS:
Other: Quality of life — Dermatology Life Quality Index, Angioedema Quality of Life Questionnaire, Angioedema Activity Score

SUMMARY:
This study aims to describe quality of life in hereditary or acquired non drug-related bradykinin-mediated angioedema patients, using validated questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Clinically documented angioedema due to C1 inhibitor deficiency, hereditary (type I et II) or acquired
* Clinically documented angioedema with normal C1 inhibitor activity (hereditary type III)

Exclusion Criteria:

* Acquired angioedema with normal C1 inhibitor activity (former "drug-induced")
* Minor subjects
* Vulnerable subjects (under guardianship/curatorship/tutorship)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hereditary or Acquired non drug-induced bradykinin-mediated angioedema patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

PRIMARY OUTCOMES:
Dermatology Life Quality Index (DLQI) | 6 months
  Description of Quality of Life (QoL) using DLQI
Angioedema Quality of Life (AE-QoL) Questionnaire | 6 months
  Description of QoL using AE-QOL questionnnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Besançon, Besançon, France